CLINICAL TRIAL: NCT03125902
Title: A Phase III, Multicenter, Randomised, Double-Blind, Placebo-Controlled Study of Atezolizumab (Anti-Pd-L1 Antibody) in Combination With Paclitaxel Compared With Placebo With Paclitaxel for Patients With Previously Untreated Inoperable Locally Advanced or Metastatic Triple Negative Breast Cancer
Brief Title: A Study of Atezolizumab and Paclitaxel Versus Placebo and Paclitaxel in Participants With Previously Untreated Locally Advanced or Metastatic Triple Negative Breast Cancer (TNBC)
Acronym: IMpassion131
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO39196; 2016-004024-29 (EudraCT Number)
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Sponsor and its agents; the study site personnel, including the investigator; and the participant will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo and Paclitaxel (Placebo Comparator): Participants will receive placebo matching to atezolizumab via IV infusion on Days 1 and 15 (± 3 days) of every 28-day cycle along with paclitaxel administered at a dose of 90 mg/m^2 via IV infusion on Days 1, 8, and 15 of every 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-PDL1 antibody; Drug: Paclitaxel
- Atezolizumab and Paclitaxel (Experimental): Participants will receive atezolizumab at a dose of 840 milligrams (mg) via intravenous (IV) infusion on Days 1 and 15 (± 3 days) of every 28-day cycle along with paclitaxel administered at a dose of 90 mg per square meter (mg/m^2) via IV infusion on Days 1, 8, and 15 of every 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-PDL1 antibody — Atezolizumab will be administered at a dose of 840 mg via IV infusion on Days 1 and 15 (± 3 days) of every 28-day cycle.
  Other Names: MPDL3280A, TECENTRIQ
  Arms: Placebo and Paclitaxel
Drug: Atezolizumab Placebo — Placebo matching to atezolizumab will be administered via IV infusion on Days 1 and 15 (± 3 days) of every 28-day cycle.
  Arms: Atezolizumab and Paclitaxel
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 90 mg/m^2 via IV infusion on Days 1, 8, and 15 of every 28-day cycle.

SUMMARY:
This Phase 3, multicenter, randomized, double-blind, placebo controlled study is designed to evaluate the efficacy and safety of atezolizumab (MPDL3280A, an anti-programmed death-ligand 1 [PD-L1] antibody) administered in combination with paclitaxel compared with placebo in combination with paclitaxel in participants with previously untreated, inoperable locally advanced or metastatic, centrally confirmed TNBC. Participants will be randomized in a 2:1 ratio to receive atezolizumab or placebo plus paclitaxel until disease progression or unacceptable toxicity or end of study, whichever occurs first (maximum up to approximately 40 months). In addition, the Sponsor may decide to terminate the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced or metastatic, histologically documented TNBC (absence of human epidermal growth factor receptor 2 [HER2], estrogen receptor [ER], and progesterone receptor [PR] expression), not amenable to surgical therapy
* Participants eligible for taxane monotherapy
* No prior chemotherapy or targeted systemic therapy (including endocrine therapy) for inoperable locally advanced or metastatic TNBC
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor block (preferred) or at least 17 unstained slides, collected ≤3 months prior to randomization, with an associated pathology report, if available. If a tumour sample taken within 3 months before randomisation is not available and a tumour biopsy is not clinically feasible, the primary surgical resection sample or the most recent FFPE tumour biopsy sample may be used. Of these additional options, the most recent sample should be used.
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Life expectancy at least 12 weeks
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end-organ function
* Negative human immunodeficiency virus (HIV) test at screening.
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening. The HBV DNA test will be performed only for patients who have a positive HBcAb test.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Women of child bearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study drug
* For men and women of child bearing potential: agreement to remain abstinent or use protocol defined contraceptive measures during the treatment period and for at least 5 months after the last dose of atezolizumab/placebo, or for at least 6 months after the last dose of paclitaxel

Exclusion Criteria:

* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 2 weeks prior to randomization
* Known central nervous system (CNS) disease, except for treated asymptomatic CNS metastases
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Uncontrolled tumor-related pain, or uncontrolled hypercalcemia or clinically significant (symptomatic) hypercalcemia
* Malignancies other than TNBC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer)
* Pregnant or breast-feeding women, or intending to become pregnant during the study
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease, cardiovascular disease, and presence of an abnormal electrocardiogram (ECG)
* Serious infection requiring antibiotics within 2 weeks prior to randomization, including but not limited to infections requiring hospitalization or IV antibiotics, such as bacteremia, or severe pneumonia
* Major surgical procedure within 4 weeks prior to randomization or anticipation of the need for a major surgical procedure during the study other than for diagnosis
* Treatment with investigational therapy within 30 days prior to initiation of study treatment
* History of hypersensitivity reactions to study drug or any component of the study drug formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2023-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (161):
- United States (8):
  - Stanford Cancer Center, Stanford, California
  - Florida Cancer Specialists; Department of Oncology, Fort Myers, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - HCA Midwest Health, Kansas City, Missouri
  - The Valley Hospital, Paramus, New Jersey
  - Magee-Woman's Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology; Sarah Cannon Research Institute, Nashville, Tennessee
- Centro Oncologico Riojano Integral (CORI), La Rioja, Argentina
- Brazil (6):
  - Centro de Pesquisas Clinicas em Oncologia - CPCO, Cachoeiro de Itapemirim, Espírito Santo
  - Santa Casa de Misericordia de Salvador, Salvador, Estado de Bahia
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Perola Byington, São Paulo, São Paulo
- Canada (9):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Kingston General Hospital, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - McGill University; Glen Site; Oncology, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke - Hopital Fleurimont, Sherbrooke, Quebec
- China (17):
  - Cancer Hospital Chinese Academy of Medical Sciences., Beijing
  - Beijing Union Hospital, Beijing
  - West China Hospital, Sichuan University; Department of Breast, Chengdu
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning cancer Hospital & Institute, Shenyang
  - Hebei Medical University Fourth Hospital;(Tumor Hospital of Hebei Province), Shijiazhuang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - The Second Affiliated Hospital of Xi'an Jiao Tong University, Xi'an
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (4):
  - Fakultni Nemocnice Hradec Kralove; Dept of Radiotherapy & Oncology, Hradec Králové
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Fakultni nemocnice Ostrava; Klinika onkologicka FNO a LF OU, Ostrava-Poruba
  - Fakultni Poliklinika Vseobecne Fakultni Niemocnice; Onkologicka Klinika, Prague
- France (17):
  - Clinique Sainte Catherine; Hopital De Semaine, Avignon
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital Morvan, Brest
  - CHD Les Oudairies, La Roche-sur-Yon
  - Centre Oscar Lambret; Senologie, Lille
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Hopital Caremeau; Hematologie Oncologie, Nîmes
  - Hopital Tenon, Paris
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Louis, Service D Oncologie Medicale, Paris
  - Ch Pitie Salpetriere; Oncologie Medicale, Paris
  - Centre Eugene Marquis; Service d'oncologie, Rennes
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Institut Gustave Roussy; Sitep, Villejuif
- Germany (13):
  - Ambulantes Tumorzentrum Spandau; Dres. Benno Mohr und Uwe Peters, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - St. Elisabeth Krankenhaus Köln GmbH; Gynäkologie und Geburtshilfe, Cologne
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - HOPA im Struensee-Haus, Dres. Erik Engel, Wiebke Hollburg, Hamburg
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz
  - OnkoNet Marburg GmbH, Marburg
  - Klinik & Poliklinik für Frauenheilkunde und Geburtshilfe, Campus Innenstadt, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Klinikum Ernst von Bergmann; Frauenklinik, Potsdam
  - Dres. Helmut Forstbauer, Carsten Ziske und Kollegen; Onkologische Schwerpunktpraxis, Troisdorf
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
- Greece (4):
  - Anticancer Hospital Ag. Savas ; 2Nd Dept. of Oncology - Internal Medicine, Athens
  - ARETAIEION UNIVERSITY HOSPITAL; oncology unit, Athens
  - Agioi Anargyroi Cancer Hospital; 2Nd Oncology Dept., Kifissia
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- India (12):
  - Yashoda Hospital, Hyderabad, Andhra Pradesh
  - Manipal Hospital; Department of Oncology, Bangalore, Karnataka
  - Tata Memorial Hospital; Dept of Medical Oncology, Mumbai, Maharashtra
  - Jehangir Hospital, Pune, Maharashtra
  - Dr. B L Kapur Memorial Hospital; BLK Cancer Centre, New Delhi, National Capital Territory of Delhi
  - Indraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Inst.&Research Center; Medical Oncology, New Delhi, National Capital Territory of Delhi
  - Max Super Speciality Hospital; Medical Oncology, North WEST Delhi, National Capital Territory of Delhi
  - Apollo Speciality Hospital, Chennai, Tamil Nadu
  - Apollo Gleneagles Hospitals, Kolkata, West Bengal
  - TATA Medical Centre; Medical Oncology, Kolkata, West Bengal
  - MAX Balaji Hospital, Delhi
- Israel (7):
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Rabin MC; Davidof Center - Oncology Institute, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Rambam Health Corporation; Oncology Institute, Rambam
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Ctr; Oncology, Tel Aviv
  - Assaf Harofeh; Oncology, Ẕerifin
- Italy (20):
  - Fondazione Università G. D'Annunzio; Clinical Research Center (CRC); Centro Studi (CESI), Chieti, Abruzzo
  - Presidio Ospedaliero S. Giovanni Di Dio; U.O. Di Oncologia, Frattamaggiore, Campania
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliero - Universitaria di Modena Policlinico, Modena, Emilia-Romagna
  - Universita Campus Bio-Medico di Roma (UCBM), Rome, Lazio
  - IRCCS Istituto Regina Elena (IFO); Oncologia Medica B, Rome, Lazio
  - Azienda Policlinico Umberto I, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova, Genoa, Liguria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo, Lombardy
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Hospital San Raffaele, Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - IEO Istituto Europeo di Oncologia;Divisione Oncologia Medica, Milan, Lombardy
  - IRCCS Istituto Clinico Humanitas; Oncologia, Rozzano (MI), Lombardy
  - Fondazione Del Piemonte Per L'oncologia IRCC Di Candiolo, Candiolo, Piedmont
  - Ospedale S. Vincenzo; Oncologia Medica, Taormina, Sicily
  - Azienda Ospedaliero-Universitaria Careggi; SOD Radioterapia, Florence, Tuscany
  - Ospedale Civile; Unita Operativa Di Oncologia Medica, Livorno, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto
- Japan (10):
  - Gunma Prefectural Cancer Center, Gunma
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Niigata Cancer Center Hospital, Niigata
  - Naha-nishi Clinic, Okinawa
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - The Cancer Institute Hospital of JFCR, Tokyo
- Morocco (2):
  - Centre Hospitalier Universitaire Mohamed VI; Oncologie-Hématologie, Marrakesh
  - Institut National D'oncologie Sidi Mohammed Ben Abdellah; Anatomopathologie, Rabat
- Romania (2):
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
- Russia (2):
  - Russian Oncology Research Center n.a. N.N. Blokhin, Moscow, Moscow Oblast
  - Petrov Research Inst. of Oncology, Saint Petersburg
- Saudi Arabia (3):
  - King Fahad Specialist Hospital; Oncology, Dammam
  - International Medical Center (IMC), Jeddah
  - King Fahad Medical City; Gastroentrology, Riyadh
- Slovakia (2):
  - Narodny Onkologicky Ustav; Oddelenie klinickej onkologie A, Bratislava
  - POKO Poprad; Department of Oncology, Poprad
- South Africa (3):
  - Wilgers Oncology Centre, Pretoria
  - Private Oncology Centre, Pretoria
  - Sandton Oncology Medical Group, Sandton
- Spain (5):
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Oncologia, A Coruña, LA Coruña
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Universitario de Fuenlabrada; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
- Turkey (Türkiye) (8):
  - Adana Baskent University Medical Faculty; Oncology, Adana
  - Ankara Bilkent City Hospital, Ankara
  - Uludag University Medical Faculty; Internal Medicine, Bursa
  - Dicle Uni Medical Faculty; Internal Medicine, Diyarbakır
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Izmir Ataturk Training and Research Hospital, Izmir
  - Kocaeli University Faculty of Medicine; Medical oncology, İzmit
  - Goztepe Prof.Dr. Suleyman Yalcin City Hospital; Clinical Oncology, Kadiköy
- United Kingdom (3):
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Christie Hospital, Manchester
  - Mount Vernon Cancer Centre, Northwood
- Vietnam (2):
  - K hospital, Hanoi
  - Hochiminh city oncology hospital, Hochiminh City

REFERENCES:
- [Derived] Miles D, Gligorov J, Andre F, Cameron D, Schneeweiss A, Barrios C, Xu B, Wardley A, Kaen D, Andrade L, Semiglazov V, Reinisch M, Patel S, Patre M, Morales L, Patel SL, Kaul M, Barata T, O'Shaughnessy J; IMpassion131 investigators. Primary results from IMpassion131, a double-blind, placebo-controlled, randomised phase III trial of first-line paclitaxel with or without atezolizumab for unresectable locally advanced/metastatic triple-negative breast cancer. Ann Oncol. 2021 Aug;32(8):994-1004. doi: 10.1016/j.annonc.2021.05.801. Epub 2021 Jul 1. PMID 34219000
- See also: Additional information for the IMpassion131 — https://www.pioneeringhealthcare.com/de/trials/breast-cancer-de/178/impassion131-de/
- See also: general information on clinical trials — https://www.wissen-immuntherapie.de/klinische-studien/studien-finden/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The target population included subjects with previously untreated inoperable locally advanced or metastatic TNBC.
Groups:
- Placebo + Paclitaxel: Participants will receive placebo matching to atezolizumab via IV infusion on Days 1 and 15 (± 3 days) of every 28-day cycle along with paclitaxel administered at a dose of 90 mg/m^2 via IV infusion on Days 1, 8, and 15 of every 28-day cycle until disease progression or unacceptable toxicity.
- Atezolizumab + Paclitaxel: Participants will receive atezolizumab at a dose of 840 milligrams (mg) via intravenous (IV) infusion on Days 1 and 15 (± 3 days) of every 28-day cycle along with paclitaxel administered at a dose of 90 mg per square meter (mg/m^2) via IV infusion on Days 1, 8, and 15 of every 28-day cycle until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Placebo + Paclitaxel | Atezolizumab + Paclitaxel
Started | 220 | 431
Completed | 0 | 0
Not Completed | 220 | 431
Not completed — Adverse Event | 0 | 1
Not completed — Death | 119 | 229
Not completed — Lost to Follow-up | 4 | 13
Not completed — Other | 0 | 4
Not completed — Physician Decision | 2 | 1
Not completed — Progressive Disease | 0 | 3
Not completed — Study Terminated By Sponsor | 74 | 143
Not completed — Withdrawal by Subject | 21 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel | Total
Number analyzed (Participants) | 220 | 431 | 651
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 176 | 322 | 498
  >=65 years | 44 | 109 | 153
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (12.2) | 54.8 (12.6) | 54.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 430 | 650
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 44 | 67
  Not Hispanic or Latino | 174 | 332 | 506
  Unknown or Not Reported | 23 | 55 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 66 | 123 | 189
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 21 | 31
  White | 128 | 246 | 374
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 14 | 37 | 51

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in the Subpopulation With Programmed Death-Ligand 1 (PD-L1)-Positive Tumour Status
Description: PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Time Frame: From Day 1 to disease progression (PD) or death from any cause, assessed up to primary completion date (approximately 26 months)
Population: PD-L1-positive subpopulation: participants in the ITT population whose PD-L1 status was IC1/2/3 at the time of randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 101 | 191
Months | 5.72 [5.39 to 7.20] | 5.95 [5.62 to 7.43]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Stratified Analysis; Test type: Superiority; p = 0.2032, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.60 to 1.12]
Statistical Analysis 2: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Unstratified Analysis; Test type: Superiority; p = 0.2601, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.62 to 1.14]

2. Primary Outcome: Progression-Free Survival (PFS) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in the Intent-to-Treat (ITT) Population
Description: as for outcome 1
Time Frame: as for outcome 1
Population: ITT population: all randomized participants, whether or not the assigned study treatment was received
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 220 | 431
Months | 5.55 [5.36 to 6.51] | 5.68 [5.42 to 7.16]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Test type: Superiority — Stratified Analysis; p = 0.1343, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.70 to 1.05]
Statistical Analysis 2: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Unstratified Analysis; Test type: Superiority; p = 0.1285, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.70 to 1.05]

3. Secondary Outcome: Overall Survival (OS) in the PD-L1-Positive Subpopulation
Description: OS is defined as the time from randomization to death from any cause. Results from a pre-specified interim analysis.
Time Frame: From Day 1 to death from any cause, assessed up 36 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 101 | 191
Months | 28.29 [19.06 to NA] — Upper limit not determined due to insufficient number of participants with events | 22.05 [19.19 to 30.52]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Stratified Analysis; Test type: Superiority; p = 0.5798, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.76 to 1.64]
Statistical Analysis 2: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Unstratified Analysis; Test type: Superiority; p = 0.4035, Log Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.80 to 1.72]

4. Secondary Outcome: Overall Survival (OS) in the ITT Population
Description: OS is defined as the time from randomization to death from any cause. Results from a pre-specified interim analysis.
Time Frame: From Day 1 to death from any cause, assessed up to end of study (up to approximately 36 months)
Population: ITT population: all randomized participants, whether or not the assigned study treatment was received
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 220 | 431
Months | 22.80 [17.08 to 28.29] | 19.19 [16.59 to 22.05]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel; Stratified analysis; Test type: Superiority; p = 0.3425, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.88 to 1.43]
Statistical Analysis 2: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Unstratified Analysis; Test type: Superiority; p = 0.2166, Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.92 to 1.48]

5. Secondary Outcome: Percentage of Participants Who Are Alive at 12 and 18 Months
Time Frame: From Day 1 to death from any cause, assessed up to 12 and 18 months
Population: ITT population: all randomized participants, whether or not the assigned study treatment was received
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 220 | 431
Percentage of Participants
  12 months | 73.47 [67.44 to 79.49] | 68.86 [64.37 to 73.34]
  18 months | 56.18 [48.94 to 63.42] | 52.32 [47.15 to 57.48]

6. Secondary Outcome: Time to Deterioration (TTD) in Global Health Status/ Health Related Quality of Life (HRQoL) in the PRO Evaluable Population
Description: Deterioration in Global Health Status/HRQoL is defined as a decrease of at least 10 points on the Global Health Status /HRQoL scale (comprised of 2 items: 29 and 30) of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The 2 items use 7-point scale (1 = very poor to 7 = Excellent). Scores are averaged, transformed to 0-100 scale; where higher score=better level of functioning or greater degree of symptoms.
Time Frame: From Day 1 to deterioration, assessed up 64 months
Population: PRO-evaluable populations: participants in the ITT population with baseline PRO assessment and at least one post-baseline PRO assessment in the questionnaire of interest (European Organization for the Research and Treatment of Cancer [EORTC] Quality-of-life Questionnaire [QLQ] C30, EORTC QLQ BR-23 or FACT-G)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 205 | 384
Months | 17.35 [9.23 to NA] — Upper limit was not reached due to not sufficient number of participants with event. | 28.68 [11.99 to NA] — Upper limit was not reached due to not sufficient number of participants with event.
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Test type: Other — Stratified analysis; p = 0.6465, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.71 to 1.24]

7. Secondary Outcome: Percentage of Participants Who Are Alive Without Progression Event at Month 12 Assessed Using RECIST v1.1
Description: PD is defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Time Frame: From Day 1 to PD or death from any cause, assessed up to 12 months
Population: ITT population: all randomized participants, whether or not the assigned study treatment was received
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 220 | 431
Percentage of Participants | 16.22 [10.18 to 22.26] | 21.63 [16.74 to 26.51]

8. Secondary Outcome: Percentage of Participants With Objective Response Assessed Using RECIST v1.1 in the PD-L1-Positive Population (Confirmed, Investigator-Assessed )
Description: Objective response is defined as complete response (CR) or partial response (PR), as determined by the investigator using RECIST v1.1 criteria. CR is defined as the disappearance of all TLs and SA reduction to less than (<) 10mm for nodal TLs/ non-TLs. PR is defined as >/=30% decrease in SD of TLs, taking as reference the baseline SD. Responses were confirmed after 8 weeks if within first 12 months or after 12 weeks if later.
Time Frame: From Day 1 to PD, assessed up to primary completion date (approximately 26 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 101 | 191
Percentage of Participants | 40.6 [30.93 to 50.82] | 49.2 [41.92 to 56.53]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Test type: Other; p = 0.1526, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.87 to 2.37]

9. Secondary Outcome: Percentage of Participants With Objective Response Assessed Using RECIST v1.1 in the PD-L1-Positive Population (Unconfirmed, Investigator-Assessed)
Description: Objective response is defined as complete response (CR) or partial response (PR), as determined by the investigator using RECIST v1.1 criteria. CR is defined as the disappearance of all TLs and SA reduction to less than (<) 10mm for nodal TLs/ non-TLs. PR is defined as >/=30% decrease in SD of TLs, taking as reference the baseline SD.
Time Frame: From Day 1 to PD, assessed up to primary completion date (approximately 26 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 101 | 191
Percentage of Participants | 55.4 [45.22 to 65.34] | 63.4 [56.09 to 70.19]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Test type: Other; p = 0.1834, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.85 to 2.31]

10. Secondary Outcome: Percentage of Participants With Objective Response Assessed Using RECIST v1.1 in the Response-Evaluable Population (Confirmed, Investigator-Assessed )
Description: as for outcome 8
Time Frame: From Day 1 to PD, assessed up to primary completion date (approximately 26 months)
Population: Response-evaluable population: participants in the ITT population with measurable disease at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 219 | 431
Percentage of Participants | 32.4 [26.27 to 39.05] | 39.9 [35.25 to 44.70]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Test type: Other; p = 0.0513, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.00 to 2.02]

11. Secondary Outcome: Percentage of Participants With Objective Response Assessed Using RECIST v1.1 in the Response-Evaluable Population (Unconfirmed, Investigator-Assessed )
Description: as for outcome 9
Time Frame: From Day 1 to PD, assessed up to primary completion date (approximately 26 months)
Population: Response-evaluable population: participants in the ITT population with measurable disease at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 219 | 431
Percentage of Participants | 47.5 [40.72 to 54.33] | 53.6 [48.76 to 58.38]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Test type: Other; p = 0.1226, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.93 to 1.81]

12. Secondary Outcome: Duration of Objective Response (DOR) Assessed Using RECIST v1.1 in DOR-evaluable Population (Unconfirmed)
Description: DOR is defined as the time period from the date of initial CR or PR until the date of PD or death from any cause, whichever occurs first. CR is defined as the disappearance of all TLs and SA reduction to <10mm for nodal TLs/ non-TLs. PR is defined as >/=30% decrease in SD of TLs, taking as reference the baseline SD. PD is defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Time Frame: From objective response to PD, assessed up to primary completion date (approximately 26 months)
Population: Duration of response (DoR)-evaluable population: participants in the ITT population with measurable disease at baseline
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 104 | 231
Months | 5.45 [4.67 to 6.31] | 6.41 [5.55 to 7.39]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Test type: Other — Unstratified Analysis; p = 0.0641, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.54 to 1.02]

13. Secondary Outcome: Percentage of Participants With Clinical Benefit Assessed Using RECIST v1.1 in Response-evaluable Population
Description: Clinical benefit is defined as the achievement of CR, PR, or stable disease according to RECIST v1.1 that lasts for at least 6 months. CR is defined as the disappearance of all TLs and SA reduction to <10mm for nodal TLs/ non-TLs. PR is defined as >/=30% decrease in SD of TLs, taking as reference the baseline SD. PD is defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. Stable disease is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference smallest SD since treatment started.
Time Frame: From Day 1 to PD, assessed up to primary completion date (approximately 26 months)
Population: Clinical Benefit Rate analysis included all participants with unconfirmed PR/CR or SD of at least 6 months duration
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 219 | 431
Percentage of Participants | 49.8 [42.96 to 56.59] | 57.1 [52.25 to 61.80]

14. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Atezolizumab in PK Evaluable Population
Time Frame: Pre-dose (0 hours) on Day 1 of Cycles 2-4 and at treatment discontinuation (TD), (approximately 9 months).
Population: PK-evaluable population: all participants who received any dose of Atezolizumab and who have at least one evaluable post-baseline PK sample. For all safety, PK and immunogenicity analyses, participants were grouped according to the treatment actually received, including cases in which atezolizumab was received in error.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 342
μg/mL
  C2D1 predose: number analyzed (Participants) | 316
  C2D1 predose | 139 (53.3)
  C3D1 predose: number analyzed (Participants) | 277
  C3D1 predose | 208 (78.3)
  C4D1 predose: number analyzed (Participants) | 243
  C4D1 predose | 242 (84.8)

15. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Atezolizumab in PK-evaluable Population
Time Frame: C1D1 30 min postdose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 308
μg/mL | 321 (90.5)

16. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Paclitaxel
Time Frame: Pre-dose (0 hours) on Day 1 of Cycle 3 (1 Cycle = 28 days)
Population: PK-evaluable population: first 60 participants who received any dose of Paclitaxel and who have at least one evaluable post-baseline PK sample. For all safety, PK and immunogenicity analyses, participants were grouped according to the treatment actually received, including cases in which atezolizumab was received in error.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 18 | 29
ng/mL | 1.51 (NA) — Insufficient number of samples analyzed. | 1.67 (NA) — Insufficient number of samples analyzed.

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Paclitaxel
Time Frame: Pre-dose (0 hours), 5-10 min before and after paclitaxel infusion, 60 min after paclitaxel infusion on Day 1 of Cycles 1 and 3 (paclitaxel infusion duration= 60 min) (1 Cycle = 28 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 23 | 36
ng/mL
  C1D1 Post-Dose | 518 (290.7) | 301 (1501)
  C3D1 Post-Dose: number analyzed (Participants) | 16 | 26
  C3D1 Post-Dose | 666 (339) | 276 (1360)

18. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: Investigator text for AEs is coded using MedDRA version 25.1
Time Frame: From Day 1 From baseline up to 64 months
Population: Safety-evaluable population: participants who received any amount of any study drug. For all safety, PK and immunogenicity analyses, participants were grouped according to the treatment actually received, including cases in which atezolizumab was received in error.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 217 | 432
Percentage of participants
  Percentage of participants with at least one AE | 97.7 | 99.1
  Percentage of participants with at least one SAE | 18.4 | 25.9

19. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies' (ADAs) Against Atezolizumab in ADA Evaluable Population
Time Frame: Pre-dose (0 hours) on Day 1 of Cycles 1, 2, 3, 4, 8, 12, 16, and at every 8 cycles thereafter until TD, at TD, and at 90-150 days after TD (maximum up to 45 months) (1 Cycle = 28 days)
Population: Anti-Drug Antibody (ADA) population:
  * Baseline ADA-evaluable population: all participants with at least one evaluable ADA assay result from a baseline sample
  * Post baseline ADA-Evaluable population: all participants with at least one evaluable ADA assay result from at least one post-baseline sample.
  For all safety, PK and immunogenicity analyses, participants were grouped according to the treatment actually received, including cases in which atezolizumab was received in error.
Measure: Number; unit: Percentage of Participants
Arm/Group | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 334
Percentage of Participants
  Percentage of participants positive for ADA at Baseline | 1.5
  Percentage of participants positive for ADA Post-baseline | 14.7

20. Secondary Outcome: Overall Survival by PD-L1 Status, Intent to Treat Population
Time Frame: From Day 1 up to 66 months
Population: ITT population: all randomized participants, whether or not the assigned study treatment was received
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 220 | 431
Months
  PD-L1 IC0: number analyzed (Participants) | 119 | 240
  PD-L1 IC0 | 20.30 [14.72 to 25.10] | 16.30 [14.52 to 19.65]
  PD-L1 IC1/2/3: number analyzed (Participants) | 101 | 191
  PD-L1 IC1/2/3 | 28.29 [19.06 to NA] — Upper limit not determined due to insufficient number of participants with events | 22.05 [19.19 to 30.52]

21. Secondary Outcome: Progression Free Survival by PD-L1 Status, Intent to Treat Population
Time Frame: From Day 1 up to primary completion date (approximately 26 months)
Population: ITT population: all randomized participants, whether or not the assigned study treatment was received
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 220 | 431
Months
  PD-L1 IC0: number analyzed (Participants) | 119 | 240
  PD-L1 IC0 | 5.49 [3.84 to 6.51] | 5.45 [4.60 to 6.51]
  PD-L1 IC1/2/3: number analyzed (Participants) | 101 | 191
  PD-L1 IC1/2/3 | 5.72 [5.39 to 7.20] | 5.95 [5.62 to 7.43]

22. Secondary Outcome: Duration of Confirmed Response (C-DoR) in (C-DoR)-Evaluable Population
Description: C-DoR is defined as the time from the first occurrence of a documented confirmed response (CR or PR) in C-DOR evaluable population until the date of disease progression per RECIST v1.1 or death from any cause, whichever occurs first. Responses were confirmed after 8 weeks if within first 12 months or after 12 weeks if later.
Time Frame: From objective response to PD, assessed up to primary completion date (approximately 26 months)
Population: Duration of confirmed response (C-DoR)-evaluable population: participants in the ITT population with measurable disease at baseline and with a confirmed objective response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo and Paclitaxel | Atezolizumab and Paclitaxel
Number analyzed (Participants) | 71 | 172
Months | 5.75 [5.36 to 7.56] | 7.66 [7.16 to 11.33]
Statistical Analysis 1: Comparison: Placebo and Paclitaxel vs Atezolizumab and Paclitaxel; Unstratified Analysis; Test type: Superiority; p = 0.01227, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.42 to 0.90]

ADVERSE EVENTS:
Time Frame: From baseline up to 64 months
Arm/Group | Atezolizumab + Paclitaxel | Placebo + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 229/431 | 119/220
Serious Adverse Events (participants affected / at risk) | 112/431 | 40/220
Other Adverse Events (participants affected / at risk) | 421/431 | 209/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Atezolizumab + Paclitaxel (N=431) | Placebo + Paclitaxel (N=220)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
BICYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 1/217 (1)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1/217 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HYPOPHYSITIS (Endocrine disorders) | 0 (0) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
KERATITIS (Eye disorders) | 1 (1) | 0 (0)
ORBITAL MYOSITIS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
IMMUNE-MEDIATED PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 2 (3) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3) | 3 (3)
DEATH (General disorders) | 4 (4) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 4 (4) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 2 (2)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
MYELITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 11 (11) | 4 (4)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 4 (4) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (4) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 2 (2) | 3 (3)
VESTIBULAR NEURONITIS (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
PROCEDURAL PNEUMOTHORAX (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPERAMYLASAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERLIPASAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POLYMYOSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBRAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
MYASTHENIA GRAVIS (Nervous system disorders) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
DEVICE BREAKAGE (Product Issues) | 1 (1) | 0 (0)
DEVICE KINK (Product Issues) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 0 (0)
GLOMERULONEPHRITIS CHRONIC (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (2) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 1 (1) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
MYELOSUPPRESSION (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 (1) | 0/217 (0)
AUTOIMMUNE PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1)
HYPOMANIA (Psychiatric disorders) | 0 (0) | 1 (1)
EMBOLISM VENOUS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atezolizumab + Paclitaxel (N=431) | Placebo + Paclitaxel (N=220)
ANAEMIA (Blood and lymphatic system disorders) | 128 (277) | 66 (134)
LEUKOPENIA (Blood and lymphatic system disorders) | 56 (181) | 20 (44)
NEUTROPENIA (Blood and lymphatic system disorders) | 98 (253) | 48 (103)
HYPERTHYROIDISM (Endocrine disorders) | 25 (28) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 49 (65) | 6 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 37 (45) | 19 (21)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 42 (47) | 15 (22)
CONSTIPATION (Gastrointestinal disorders) | 82 (103) | 33 (56)
DIARRHOEA (Gastrointestinal disorders) | 130 (209) | 50 (88)
DRY MOUTH (Gastrointestinal disorders) | 24 (32) | 8 (9)
DYSPEPSIA (Gastrointestinal disorders) | 17 (18) | 11 (12)
NAUSEA (Gastrointestinal disorders) | 117 (167) | 54 (108)
STOMATITIS (Gastrointestinal disorders) | 23 (29) | 10 (18)
VOMITING (Gastrointestinal disorders) | 70 (110) | 20 (36)
ASTHENIA (General disorders) | 101 (149) | 47 (61)
FATIGUE (General disorders) | 119 (154) | 57 (73)
OEDEMA PERIPHERAL (General disorders) | 52 (66) | 22 (29)
PYREXIA (General disorders) | 68 (92) | 25 (39)
NASOPHARYNGITIS (Infections and infestations) | 34 (41) | 16 (19)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 29 (45) | 18 (22)
URINARY TRACT INFECTION (Infections and infestations) | 36 (48) | 11 (15)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 86 (168) | 38 (62)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 87 (165) | 39 (68)
NEUTROPHIL COUNT DECREASED (Investigations) | 68 (361) | 35 (220)
WEIGHT DECREASED (Investigations) | 32 (35) | 6 (6)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 65 (285) | 30 (203)
DECREASED APPETITE (Metabolism and nutrition disorders) | 66 (106) | 22 (33)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 69 (96) | 21 (25)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 40 (51) | 20 (23)
MYALGIA (Musculoskeletal and connective tissue disorders) | 48 (59) | 25 (34)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 48 (61) | 23 (34)
DIZZINESS (Nervous system disorders) | 38 (43) | 20 (23)
DYSGEUSIA (Nervous system disorders) | 36 (39) | 16 (19)
HEADACHE (Nervous system disorders) | 59 (76) | 38 (44)
HYPOAESTHESIA (Nervous system disorders) | 26 (37) | 16 (20)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 126 (173) | 60 (83)
PARAESTHESIA (Nervous system disorders) | 40 (52) | 22 (30)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 44 (52) | 23 (26)
INSOMNIA (Psychiatric disorders) | 33 (40) | 22 (22)
BREAST PAIN (Reproductive system and breast disorders) | 28 (34) | 9 (10)
COUGH (Respiratory, thoracic and mediastinal disorders) | 86 (109) | 37 (44)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 49 (57) | 24 (29)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 26 (30) | 15 (18)
ALOPECIA (Skin and subcutaneous tissue disorders) | 253 (257) | 118 (124)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 25 (29) | 8 (8)
PRURITUS (Skin and subcutaneous tissue disorders) | 47 (74) | 19 (22)
RASH (Skin and subcutaneous tissue disorders) | 78 (108) | 36 (51)
HOT FLUSH (Vascular disorders) | 19 (21) | 11 (12)
HYPERTENSION (Vascular disorders) | 20 (35) | 12 (13)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 22 (41) | 9 (21)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 22 (32) | 6 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/02/NCT03125902/Prot_001.pdf
  • Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT03125902/SAP_000.pdf